CLINICAL TRIAL: NCT03552081
Title: Tobacco and Sperm Genome: Effects of Smoking Cessation
Acronym: TABAGERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0344
Record Dates: First submitted 2018-04-25; First posted 2018-06-11 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Male Infertility
Keywords: spermatogenesis; tobacco; DNA Fragmentation Index
MeSH Terms: conditions — Infertility, Male | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fragmented DNA evaluation in blood and semen samples (Experimental): 20 men followed for smoking cessation will be included in the study in order to evaluate the time required for the repair of the sperm abnormalities and in particular the DNA of the gametes generated by the smoking
  Interventions: Other: Fragmented DNA evaluation in blood and semen samples

INTERVENTIONS:
Other: Fragmented DNA evaluation in blood and semen samples — The objective will be to evaluate the decrease in the percentage of sperm with spermatic DNA fragmentation by the TUNEL technique following the evolution of this rate to 3 months, 6 months and 12 months after cessation of smoking by blood and semen samples.

SUMMARY:
Tobacco is a male infertility risk factor. Many studies comparing smokers to non-smokers have shown effects on spermatogenesis and the quality of the male gamete. In vitro fertilization success rates are decreased in smokers and in natural procreation the time required to conceive (excellent fertility indicator) seems to be lengthened in the smoker. The prospective study that the investigators propose to carry out would make it possible to know the time required for the repair of the sperm abnormalities and in particular the DNA of the gametes generated by the smoking.

DETAILED DESCRIPTION:
Tobacco is a male infertility risk factor. Many studies comparing smokers to non-smokers have shown effects on spermatogenesis and the quality of the male gamete. In vitro fertilization success rates are decreased in smokers and in natural procreation the time required to conceive (excellent fertility indicator) seems to be lengthened in the smoker. Tobacco is a well-known mutagen. It will induce damage to the male gametes DNA. Tobacco increases the oxydation of DNA. Exposure to tobacco increases the percentage of spermatozoa with broken DNA or defective chromatin and induces gametes aneuploidy as has been reported in several studies. The set of effects of tobacco on the male gametes questions the consequences for the conceptus (from embryo to adult). The prospective study that the investigators propose to carry out would make it possible to know the time required for the repair of the sperm abnormalities and in particular the DNA of the gametes generated by the smoking. Indeed, a cycle of spermatogenesis extending over 74 days, it would be important to know if it is necessary to wait a complete cycle or even more before proposing a management. It would therefore be possible to find the most favorable period for reducing tobacco-related risks and for effective management.

A blood test will be performed at T0 (before weaning) and during follow-up at 3, 6 and 12 months for the determination of the Inhibin hormones and testosterone. Sperm analysis at the different follow-up times will be carried out at CECOS using a standardized methodology (WHO). Two tests of analysis will be used in this study on each sample: the TUNEL test and the SCSA. A measurement of DNA oxidation will also be performed, as well as a study of spermatic aneuploidy (in situ hybridization technique of fluorescent centromeric chromosomal probes).

ELIGIBILITY:
Inclusion Criteria:

* 1st Consultation in the Tobacco Control Co-ordination Unit,
* Affiliate or beneficiary of a social security scheme
* Free, informed and written consent signed by the participant and the investigator

Exclusion Criteria:

* febrile state during the 3 months before inclusion,
* antecedent consultation for male infertility,
* BMI> 30,
* Medical and / or surgical history that can alter spermatogenesis -Chemotherapy / Radiation Therapy / IRA-therapy, Cryptorchidism, testicular Torsion, significant varicocele, chronic, progressive disease,
* hypovolemia <1.6ml
* Major persons protected by law (guardianship, curators, safeguarding of justice)
* Patients in periods of exclusion for another clinical research protocol
* Co-addiction (cannabis, alcohol, other drugs)
* Neuropsychiatric Pathology, considered serious by the investigator
* Psychotropic treatment (antidepressant, anxiolytic, antipsychotic)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Change of the Percentage of spermatozoa presenting a fragmented DNA from Baseline to 12 months after smoking cessation | Up to 12 months after smoking cessation
  TUNEL technique will be performed to evaluate the percentage of spermatozoa presenting a fragmented DNA at day 0 (before weaning = baseline), and 12 months after smoking cessation
Change of the Percentage of spermatozoa presenting a fragmented DNA from Baseline to 3 months after smoking cessation | Up to 3 months after smoking cessation
  TUNEL technique will be performed to evaluate the percentage of spermatozoa presenting a fragmented DNA at day 0 (before weaning = baseline), and 3 months after smoking cessation
Change of the Percentage of spermatozoa presenting a fragmented DNA from Baseline to 6 months after smoking cessation | Up to 6 months after smoking cessation
  TUNEL technique will be performed to evaluate the percentage of spermatozoa presenting a fragmented DNA at day 0 (before weaning = baseline), and 6 months after smoking cessation

SECONDARY OUTCOMES:
Rate of 8-OHdG gamete DNA | Up to 12 months after smoking cessation
Spermogram exam | Up to 12 months after smoking cessation
  Spermogram examination
Fragmentation index (DFI) of gamete DNA | Up to 12 months after smoking cessation
Aneuploid sperm count | Up to 12 months after smoking cessation
luteinizing hormone (LH) levels luteinizing hormone (LH) levels luteinizing hormone (LH) levels | Up to 12 months after smoking cessation
  Blood samples at day 0 (before weaning), and at 3 months, 6 months, 12 months after smoking cessation
Testosterone levels | Up to 12 months after smoking cessation
  Blood samples at day 0 (before weaning), and at 3 months, 6 months, 12 months after smoking cessation

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Moreau, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Service de médecine de la reproduction, Toulouse, France